CLINICAL TRIAL: NCT01104428
Title: Research on the Blood- Cooling - Toxin - Removing - Stasis - Dispersing Protocol Evaluation of Hench-schonlein Purpura
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaoning University of Traditional Chinese Medicine (Other)
Collaborators: Dongzhimen Hospital, Beijing (Other); Shenyang Hospital of Integrated Traditional and westen Medicine (Unknown); Dalian Children's Hospital (Other)
Responsible Party: President Guanlin Yang, Affiliated Hospital of Liaoning University of Traditional Chinese Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: zhangjun555678
Record Dates: First submitted 2010-01-25; First posted 2010-04-15 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Purpura, Schoenlein-Henoch
Keywords: Hench-schonlein purpura; Renal damage; Relapse; End event; TCM syndrome
MeSH Terms: conditions — IgA Vasculitis; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Drug:"ziying" (Experimental)
  Interventions: Drug: "ziying" granules

INTERVENTIONS:
Drug: Placebo — granules, <10years,10g,Three times a day,take orally >10years,20g,Three times a day,take orally fore weeks a period,Observe 2 periods
  Arms: placebo
Drug: "ziying" granules — granules, <10years,10g,Three times a day,take orally >10years,20g,Three times a day,take orally fore weeks a period,Observe 2 periods
  Arms: Drug:"ziying"

SUMMARY:
Due to high incidence of renal damage by Hench-schonlein Purpura(HSP) is the key to affect prognosis, this project moves the research emphasis forward in line with the idea of "prevention of progress of disease", Which concerns on Traditional Chinese Medicine(TCM) clinical research scheme evaluation of HSP, evaluates the renal damage and disease recurrence as the end event, and comes to the evaluation through the comparative study that the vantage point of the scheme of syndrome differentiation and treatment in detoxification, cooling blood and removing blood stasis to the conventional treatments can reduce kidney damage and recurrence rate.

DETAILED DESCRIPTION:
Target：Optimize the TCM scheme of syndrome differentiation and treatment of HSP in line with the idea of blood- Cooling - Toxin - Removing - Stasis - Dispersing under the path of combination between disease differentiation and syndrome differentiation, and regards reducing the rate of the recurrence of HSP and kidney damage as the end point of evaluation indexes, to evaluate the clinical efficacy of the scheme scientifically. Main research contents: Retrospective case investigation, analysis and research on literature, research on clinical assessment of the scheme of syndrome differentiation and treatment. Methods：With a series of compounds as the main interference factors, choosing the sample estimation of superiority design and adopting the test methods of randomized, double-blind, placebo-controlled to carry out the research of multicenter clinical efficacy evaluation.

It summarizes the advantages and rules of syndrome differentiation and treatment in TCM by means of the comparative study, which provides technical guidelines for the industry and sets an example to summarize the key common technology of clinical research, and also improves the evaluation level of TCM clinical research and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* To comply with the diagnostic standard of purpura in TCM and Hench-schonlein purpura in western medicine;
* To comply with the diagnostic standard of TCM syndrome differentiation;
* Age between 5 and 18;
* without similar herbal treatment a week before being included;
* Informed Consent Form is required to be singed.

Exclusion Criteria:

* Fall short of the diagnostic standard of purpura in TCM and Hench-schonlein purpura in western medicine;
* Fall short of the diagnostic standard of TCM syndrome differentiation;
* Older then 18 years or younger then 5years;
* Take similar herbal treatment within a week before being included;
* Can not take the drug according to the regulation or follow-up on time
* Patients combine serious primary disease in respiratory、gastrointestinal、hemopoietic、renal，or psychosis,or pestilence;
* Allergic to drugs of this research or others;
* human subject of other clinical research in the nearly tow weeks.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 256 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
whether endpoint such as renal damage or disease recurrence appears in the participants. | 6 months
  Endpoint is a mark of termination or completion. In this clinical research, the renal damage and disease recurrence that constitutes the target outcomes of the trial.

SECONDARY OUTCOMES:
whether the TCM syndrome of participants disappears after treatment. | 1 month
  Optimize the TCM scheme of syndrome differentiation and treatment of HSP in line with the idea of blood- Cooling - Toxin - Removing - Stasis - Dispersing, under the path of combination between disease differentiation and syndrome differentiation In the process of disease of a series of function, metabolism and morphological structure changes caused by the subjective feeling of abnormal patient as symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: zhang jun, master, Study Chair — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; zhao lijun, master, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; wang shaojie, master, Principal Investigator — Dalian Children's Hospital; ma liming, master, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; li tienan, master, Principal Investigator — Shenyang Hospital of Integrated Traditional and westen Medicine; xu rongqian, master, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Zhangjun, Shenyang, Liaoning, China